CLINICAL TRIAL: NCT01267240
Title: A Phase II Study of Vorinostat and Capecitabine in Recurrent and/or Metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN) and Nasopharyngeal Carcinoma (NPC)
Brief Title: Capecitabine and Vorinostat in Treating Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study treatment did not show clinical activity.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02556; NCI-2011-02556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMH-PHL-068; CDR0000689859; NCI 8192; PHL-068 (Other: University Health Network-Princess Margaret Hospital); 8192 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH)
Record Dates: First submitted 2010-12-24; First posted 2010-12-28 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Paranasal Sinus Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage IVA Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Hypopharyngeal Squamous Cell Carcinoma; Stage IVB Laryngeal Squamous Cell Carcinoma; Stage IVB Oral Cavity Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Hypopharyngeal Squamous Cell Carcinoma; Stage IVC Laryngeal Squamous Cell Carcinoma; Stage IVC Oral Cavity Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (capecitabine, vorinostat) (Experimental): Patients receive capecitabine PO BID and vorinostat PO daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Vorinostat

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This partially randomized phase II trial studies giving capecitabine and vorinostat in treating patients with head and neck cancer that has come back after previous treatment or that has spread to other areas in the body. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving capecitabine together with vorinostat is more effective than capecitabine alone in treating patients with cancer of the head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate (complete and partial) and duration of response of the combination of vorinostat and capecitabine in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN). (SCCHN) II. To determine the objective response rate (complete and partial) and duration of response of the combination of vorinostat and capecitabine in patients with recurrent and/or metastatic nasopharyngeal carcinoma (NPC). (NPC)

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of vorinostat and capecitabine in patients with recurrent and/or metastatic SCCHN. (SCCHN) II. To determine the rate of progression-free survival (PFS) at 6 months. (SCCHN) III. To determine the rate and duration of stable disease (SD). (SCCHN) IV. To determine the median PFS, and the rate of PFS at 1 year. (SCCHN) V. To determine the median overall survival (OS), and rates of overall survival at 6 months and at 1 year. (SCCHN) VI. To evaluate the safety and tolerability of the combination of vorinostat and capecitabine in patients with recurrent and/or metastatic NPC. (NPC) VII. To determine the duration of objective response. (NPC) VIII. To determine the rate and duration of stable disease (SD). (NPC) IX. To determine the median PFS, and the rate of PFS at 1 year. (NPC) X. To determine the median overall survival (OS), and rates of overall survival at 6 months and at 1 year. (NPC)

OUTLINE: This is a non-randomized, open-label study of patients with SCCHN and NPC (Stage I), followed by a randomized study of patients with NPC (Stage II).

STAGE I: Patients receive capecitabine orally (PO) twice daily (BID) and vorinostat PO daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

STAGE II: Patients with NPC are randomized to 1 of 2 treatment arms.

ARM I: Patients receive capecitabine PO BID and vorinostat PO daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients will be followed up at 3-4 weeks and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed SCCHN or NPC that is recurrent and/or metastatic and that is not amendable to curative therapy by surgery or radiation; SCCHN originating from the following sites are eligible: oral cavity, oropharynx, larynx, hypopharynx and paranasal sinus are eligible; for patients with a diagnosis of SCCHN of unknown origin, their eligibility must be reviewed and approved by the principal investigator
* For patients with SCCHN, they may have received one prior targeted therapy for recurrent or metastatic disease (excluding histone deacetylase [HDAC] inhibitors) provided treatment is completed > 4 weeks prior to enrollment; they may have received prior systemic chemotherapy (ie, induction, concurrent or adjuvant) for SCCHN as part of the initial multimodality treatment for locally advanced disease if the chemotherapy is completed > 6 months prior to enrollment; patients are not eligible if they received fluorouracil (5-FU) or capecitabine previously as part of the initial multimodality treatment
* Patients with NPC must have completed one prior chemotherapy regimen for recurrent or metastatic disease at least 4 weeks prior to enrollment; in addition, they may have received prior systemic chemotherapy (ie, induction, concurrent or adjuvant) for NPC as part of the initial multimodality treatment for locally advanced disease if the chemotherapy is completed > 6 months prior to enrollment; patients are eligible if they received 5-FU as part of the initial multimodality treatment; patients are not eligible if they received capecitabine previously
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan; indicator lesions must not have been previously treated with surgery, radiation therapy or radiofrequency ablation unless there is documented progression after therapy
* Patients must have completed any previous surgery or radiotherapy >= 4 weeks prior to enrollment
* Previously treated patients must have evidence of progressive disease, either clinically or radiographically, as assessed by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%)
* Life expectancy of greater than 12 weeks
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.25 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN or =< 5 x ULN with documented liver metastases
* Creatinine =< 1.25 x ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above 1.25 x ULN
* 12-lead electrocardiogram (ECG) with normal tracing, or non-clinically significant changes that do not require medical intervention; corrected QT (QTc) interval < 470 msec, and without history of Torsades de Pointes or other symptomatic QTc abnormality
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity of vorinostat will be determined following review of their case by the principal investigator
* Women of childbearing potential and men must be surgically sterilized, practicing abstinence, or agree to use 2 birth control methods prior to study entry and for the duration of study participation; the 2 birth control methods can be either be 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy; the following are considered adequate barrier methods of contraception: diaphragm or sponge, and condom; other methods of contraception such as copper intrauterine device or spermicide may be used; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Willingness to discontinue taking any medications that are generally accepted to have a risk causing Torsades de Pointes during the study

Exclusion Criteria:

* Past or current malignancy other than SCCHN or NPC, except for:

  * Cervical carcinoma Stage 1B or less
  * Non-invasive basal cell and squamous cell skin carcinoma
  * Malignant melanoma with a complete response of a duration of > 10 years
  * Radically treated prostate cancer (prostatectomy or radiotherapy) with normal prostate specific antigen (PSA), and not requiring ongoing anti-androgen hormonal therapy
  * Other cancer diagnosis with a complete response of duration of > 5 years
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* Prior use of capecitabine is not allowed
* Prior and concomitant treatment with HDAC inhibitors (such as valproic acid) are not allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or other agents used in study
* Patients who are unable to take oral medications and / or who have a clinical or radiological diagnosis of bowel obstruction are ineligible
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, active peptic ulcer disease, myocardial infarction within 6 months prior to entry, congestive heart failure, symptomatic congestive heart failure, active cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat
* Human immunodeficiency virus (HIV)-positive patients are ineligible
* Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency are excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (14):
- United States (9):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Veterans Administration Hospital - Martinez, Martinez, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre-Corporate, London, Ontario
  - London Regional Cancer Program, London, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Capecitabine, Vorinostat)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (Capecitabine, Vorinostat)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Region of Enrollment [Number; unit: participants]
  Canada | 22
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate According to Response Evaluation Criteria in Solid Tumors
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT and MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Arm I (Capecitabine, Vorinostat)
Number analyzed (Participants) | 25
participants | 2

2. Secondary Outcome: Survival
Description: Overall survival is defined as the length of time from start of treatment to death from any cause. Estimated using the Kaplan-Meier method.
Time Frame: Up to 1 year
Population: 16 patients of the 25 were eligible for response assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Capecitabine, Vorinostat)
Number analyzed (Participants) | 16
months | 10.8 [5 to NA] — Not reached

3. Secondary Outcome: Progression-free Survival
Description: PFS is defined as the duration of time from start of treatment to time of progression, death, or completion of the 1-year follow-up, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: From time of treatment initiation to disease progression, death, or completion of the 1 year follow-up, whichever occurs first.
Population: 16 of 25 patients were evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Capecitabine, Vorinostat)
Number analyzed (Participants) | 16
months | 2.3 [1.2 to 3.6]

ADVERSE EVENTS:
Arm/Group | Arm I (Capecitabine, Vorinostat)
Serious Adverse Events (participants affected / at risk) | 7/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Capecitabine, Vorinostat) (N=25)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Other: diverticulitis (Gastrointestinal disorders) | 1 (1)
Ischemia cerbrovascular (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Capecitabine, Vorinostat) (N=25)
Fatigue (General disorders) | 23
Lymphocyte count decreased (Investigations) | 21
Anemia (Blood and lymphatic system disorders) | 16
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 13
Hyponatremia (Metabolism and nutrition disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Platelet count decreased (Investigations) | 10
Palmar-plantar erythrodysethesia syndrome (Skin and subcutaneous tissue disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Dysphagia (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Mucositis oral (Gastrointestinal disorders) | 10
Hypertension (Vascular disorders) | 10
Insomnia (Psychiatric disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 8
Creatinine increased (Investigations) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 7
White blood cell decreased (Investigations) | 6
Headache (Nervous system disorders) | 6
Tinnitus (Ear and labyrinth disorders) | 6
Hypothyroidism (Endocrine disorders) | 6
Anxiety (Psychiatric disorders) | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Depression (Psychiatric disorders) | 5
Edema limbs (General disorders) | 5
Proteinuria (Renal and urinary disorders) | 5
Weight loss (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Facial pain (General disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Urinary frequency (Renal and urinary disorders) | 4
Edena face (General disorders) | 4
Trismus (Musculoskeletal and connective tissue disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Confusion (Psychiatric disorders) | 3
Hypomagnesmia (Metabolism and nutrition disorders) | 3
Blood bilirubin increased (Investigations) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Neutrophil count decreased (Investigations) | 3
Ear pain (Ear and labyrinth disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 2
Dizziness (Nervous system disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Alkaline phosphatase increased (Investigations) | 2
Thromboembolic event (Vascular disorders) | 2
Aspartate amino transferase increased (Investigations) | 2
Oral pain (Gastrointestinal disorders) | 2
Dry eye (Eye disorders) | 2
Flu like symptoms (General disorders) | 2
Glucose intolerance (Metabolism and nutrition disorders) | 2
Repiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Paresthesia (Nervous system disorders) | 1
INR increased (Investigations) | 1
Agitation (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrilation (Cardiac disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Weight gain (Investigations) | 1
Cataract (Eye disorders) | 1
Somnolence (Nervous system disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Gait disturbance (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Dysarthria (Nervous system disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to lack of activity of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less